CLINICAL TRIAL: NCT03521232
Title: A Phase I/IIA, Open-Label, Three-Stage Study to Investigate the Safety, the Efficacy and the Pharmacokinetics of Niclosamide Enemas in Subjects With Active Ulcerative Proctitis or Ulcerative Procto-Sigmoiditis
Brief Title: A Study of Niclosamide Enemas in Subjects With Active Ulcerative Proctitis or Ulcerative Proctosigmoiditis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Covid-19
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FW-UC-2017
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-08

CONDITIONS: Ulcerative Colitis; Ulcerative Proctitis; Ulcerative Proctosigmoiditis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 150 mg/60 ml (Experimental): Niclosamide enemas 150 mg/60 ml given twice daily for 6 weeks
  Interventions: Drug: Niclosamide
- 450 mg/60 ml (Experimental): Niclosamide enemas 450 mg/60 ml given twice daily for 6 weeks
  Interventions: Drug: Niclosamide

INTERVENTIONS:
Drug: Niclosamide — enema given twice daily for 6 weeks

SUMMARY:
This will be a phase I/IIa, open-label, three-stage, single center study aimed at investigating the safety, the efficacy (clinical and endoscopic effects) and the pharmacokinetics of Niclosamide enema 150 mg/60 ml and 450 mg/60 ml in subjects with mild-to-moderate UP and UPS, defined as a Modified Mayo Score (MMS) ≥ 4 and < 8, with a stool frequency subscore (SFS) ≥ 1, a rectal bleeding sub-score (RBS) = 1 or 2, and an endoscopic subscore (mucosal appearance) = 1 or 2. At the endoscopic sub-score any degree of friability will be classified as having a sub-scale score of 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years at the time of signing the informed consent;
2. Must understand and voluntarily sign an informed consent from (ICF) prior to any study-related assessments/procedures being conducted.
3. Must be able to adhere to the study visit schedule and other protocol requirements;
4. Diagnosis of UP or UPS with a duration of at least 3 months prior to the Screening Visit
5. MMS score ≥4 to < 8 (range: 0-9) prior to enrolment in the study.
6. Availability to perform an endoscopy (colonoscopy or flexible rectosigmoidoscopy);

Exclusion Criteria:

1. Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, microscopic colitis, radiation colitis, or diverticular disease-associated colitis;
2. UC extended more than 40 cm from the anal verge;
3. Subjects who have had surgery as a treatment for UC or who, in the opinion of the Investigator, are likely to require surgery for UC during the study;
4. History of any clinically significant neurological, renal, hepatic, gastrointestinal, pulmonary, metabolic, psychiatric, endocrine, hematological disorder or disease or any other medical condition that, in the Investigator's opinion, would preclude participation in the study;
5. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she was to participate in the study or confounds the ability to interpret data from the study;
6. Pregnant or breast feeding females;
7. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis, atypical mycobacterial disease, and herpes zoster), human immunodeficiency virus (HIV), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) or oral antibiotics within 4 weeks of screening;
8. Subjects who have received any investigational drug or device in the last 3 months;
9. History of alcohol, drug, or chemical abuse within the last 6 months;
10. Known hypersensitivity to niclosamide or any excipients in the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Niclosamide enemas 150 mg/60 ml and 450 mg/60 ml graded according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0. | baseline to 6 weeks
  1. Number of subjects with serious adverse reactions (i.e. treatment-related) during 6 weeks of treatment with Niclosamide enemas;
  2. Number of subjects with grade ≥ 3 adverse reactions during 6 weeks of treatment with Niclosamide enemas;
  3. Number of subjects with grade ≥ 2 adverse reactions during 6 weeks of treatment with Niclosamide enemas.

SECONDARY OUTCOMES:
Number of subjects with clinical remission defined as MMS* ≤ 2 with no individual subscore >1 after 6 weeks of treatment | baseline to 6 weeks

OTHER OUTCOMES:
Change in signs and symptoms (rectal bleeding and stool frequency) from baseline to 2, 4 and 6 weeks of treatment | from baseline to 2, 4 and 6 weeks
Change in sigmoidoscopic score (mucosal appearance) from baseline to 6 weeks of treatment | baseline to 6 weeks
Change in hs-CRP and fecal calprotectin from baseline to 2, 4 and 6 weeks of treatment | baseline to 2, 4 and 6 weeks
Change in histology (Geboes index) from baseline to 6 weeks of treatment | baseline to 6 weeks
Change in safety laboratory tests from baseline to 6 weeks of treatment | baseline to 6 weeks
  the number of subjects with values low, normal, and high compared to the normal ranges pretreatment versus post-treatment will be provided
Change in 12-lead ECG parameters from baseline to 2, 4 and 6 weeks of treatment | baseline to 2, 4 and 6 weeks of treatment
  1. PR interval 2. RR interval 3. QRS interval 4 QT interval 5. HR interval 6. QtcF interval. All intervals summarized descriptively by visit
Change in heart rate from baseline to 2, 4 and 6 weeks of treatment | baseline to 2, 4 and 6 weeks
  summarized descriptively by visit and presented as shift tables
Change in quality of life (12-item Short-Form) from baseline to 6 weeks of treatment | baseline to 6 weeks
Plasma levels of niclosamide measured before and after dosing | baseline to 6 weeks
Change in sitting systolic and diastolic blood pressure from baseline to 2, 4 and 6 weeks of treatment | baseline to 2, 4 and 6 weeks
  summarized descriptively by visit and presented as shift tables
Change in body temperature from baseline to 2, 4 and 6 weeks of treatment | baseline to 2, 4 and 6 weeks
  summarized descriptively by visit and presented as shift tables

CONTACTS AND LOCATIONS:
Overall Officials: James Pennington, M.D., Study Director — First Wave BioPharma
Locations (1):
- Tor Vegata, Rome, Italy

IPD SHARING:
Plan to Share IPD: No